CLINICAL TRIAL: NCT02602119
Title: Intraoperative Imaging of Pulmonary Nodules by OTL38
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 822153; NCT02769156 (obsolete NCT alias)
Record Dates: First submitted 2015-11-02; First posted 2015-11-11 (Estimated); Last update posted 2022-06-28 (Actual); Status verified 2022-06

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms | interventions — Pafolacianine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- OTL38 (Experimental): Dosage calculated by weight of individual
  Interventions: Drug: OTL38

INTERVENTIONS:
Drug: OTL38 — Infusion of OTL38 prior to surgery

SUMMARY:
The primary end-point of the study is to determine the sensitivity of OTL in identifying lung nodules when excited by an imaging probe. Investigators intend to enroll 300 lung cancer patients in this study. The study is focusing on patients presenting with suspected malignancies of the lung and pleura who are considered to be good surgical candidates.

DETAILED DESCRIPTION:
According to the World Health Organization, lung cancer is the most common cause of cancer-related death in men and women, and is responsible for 1.5 million deaths worldwide annually as of 2012. Surgery remains the best option for patients presenting with operable Stage I or II cancers, however the five year survival rate for these candidates remains at a dismal 73% for Stage I and 53% for Stage II. The high rates of local recurrence suggest that surgeons are unable to completely detect and remove primary tumor nodules in a satisfactory manner as well as lingering metastases in sentinel lymph nodes. By ensuring a negative margin through imaging during surgery it would be possible for the investigators to improve the rates of recurrence free patients and thus overall survival.

Thoracic malignancies are the ideal disease to investigate intra-operative imaging. Over 85% of lung and pleural malignancies express folate receptor alpha (FRA), therefore making folate receptors (FR) the ideal targets for imaging agents. While folate will initially distribute to all cells, redistribution, metabolism, and excretion will eliminate most of this agent from healthy tissues within hours. Tumor cells that over express FRα will retain folate and any fluorescent labeled folate conjugate and internalize this. It is important to note that FRA is expressed only in the proximal tubules of the kidneys, activated macrophages, and in the choroidal plexus. However, the fluorescence signal in the kidneys is expected to be significantly lower than the tumor tissues. Thus, the false positive detection rate is expected to be extremely low.

The investigators have conducted a Phase I clinical trial with folate-FITC in 50 patients with lung cancer. In the study at UPenn, the investigators had no adverse events. The investigators had excellent sensitivity and specificity with this technique with only grade 1 side effects (allergic reaction). All side effects reversed when the injection was halted. This study confirmed that FRA is a reasonable target for lung cancer.

On Target Laboratories, LLC has developed OTL38. Compared with some of the existing fluorescent imaging agents, OTL38 is associated with less auto-fluorescence due to its near-IR excitation wavelength and can be seen through blood and tissues up to 1.5 cm thickness. Thus, in this study, the investigator's goal has changed from the folate-FITC formulation to the OTL38 formulation. The fluorophore component of the drug is new, whereas the target and design of the study remain unchanged.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients over 18 years of age
* Patients presenting with a lung or pleural nodule or mass presumed to be resectable on pre- operative assessment
* Good operative candidate
* Subject capable of giving informed consent and participating in the process of consent.

Exclusion Criteria:

* Pregnant women as determined by urinary or serum beta hCG within 72 hours of surgery
* Patients with a history of anaphylactic reactions to OTL38
* Patients with a known allergy to Benadryl
* At-risk patient populations:

  * Homeless patients
  * Patients with drug or alcohol dependence
  * Children and neonates
  * Patients unable to participate in the consent process.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 262 (Actual)
Dates: Start 2015-05; Primary Completion 2022-05 (Actual); Study Completion 2022-05 (Actual)

PRIMARY OUTCOMES:
Ability of the imaging system to detect the expression of the OTL38 in the nodule/mass (i.e tumor) and discern the uptake of the dye by the tumor. | 5 years
  Detected with imaging probe.
Microscopic examination and immunohistochemistry of tumor | 5 years
  Performed by a pathologist. This will allow investigators to compare pathology results with video images taken by imaging probe to calculate false positive (i.e., identification of non FRA-positive tumors) rates of OTL38.

SECONDARY OUTCOMES:
Incidence rates of all AEs, treatment-emergent adverse events (TEAEs) and adverse device events (ADEs) from time of OTL38 administration through participants' first, post-operative appointment with surgeon. | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Sunil Singhal, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States